CLINICAL TRIAL: NCT02431975
Title: Latency and Early Neonatal Provision of Antiretroviral Drugs Clinical Trial
Acronym: LEOPARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Witwatersrand, South Africa (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Louise Kuhn, Professor of Epidemiology, Department of Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO5011; U01HD080441 (NIH)
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: HIV; infant; antiretroviral therapy, highly active; antiretroviral agents
MeSH Terms: interventions — Nevirapine; Zidovudine; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early ART (Experimental): All infants enrolled in the trial, regardless of maternal PMTCT regimen, will be initiated on a triple ARV regimen consisting of nevirapine (NVP), zidovudine (ZDV) and lamivudine (3TC) presumptively based on the initial positive result. This regimen will be continued to 42 weeks post menstrual age (PMA). At this time, infants will be switched to LPV/r, ZDV and 3TC to be continued to 104 weeks or longer unless otherwise preferred by the treating clinician or if any clinical or laboratory contraindications are identified.
  Interventions: Drug: Nevirapine; Drug: Zidovudine; Drug: Lamivudine; Drug: LPV/r

INTERVENTIONS:
Drug: Nevirapine — Standard medication used to treat and prevent HIV/AIDS, specifically HIV-1. It is generally recommended for use with other antiretroviral medication.
  The initial dose of NVP will be 6 mg per kg per dose orally twice daily until 42 weeks gestational age (2 weeks of age for infants born at term) which is the dosing selected by the NIH International Maternal, Pediatric, Adolescent AIDS Clinical Trials (IMPAACT) Network.
  Other Names: NVP; Viramune
Drug: Zidovudine — An antiretroviral medication used to prevent and treat HIV/AIDS. It is generally recommended for use with other antiretroviral.
  ZDV will be dosed as per standard guideline and routine practices.
  Other Names: ZDV; Retrovir
Drug: Lamivudine — An antiretroviral medication used to prevent and treat HIV/AIDS. It is effective against both HIV-1 and HIV-2.
  3TC will be dosed as per standard guideline and routine practices.
  Other Names: 3TC; Epivir
Drug: LPV/r — Lopinavir is an antiretroviral of the protease inhibitor class. It is used against HIV infections as a fixed-dose combination with another protease inhibitor, ritonavir.
  LPV/r will be dosed as per standard guideline and routine practices.
  Other Names: Ritonavir-boosted lopinavir

SUMMARY:
The investigators propose a non-randomized clinical trial of 60 HIV-infected infants identified within 48 hours of birth and their mothers to investigate the consequences of very early ART on the establishment and maintenance of the viral reservoir.

The first phase (early ART initiation within 48 hours of birth) will examine the trajectory i.e. changes over time of the viral reservoir and detection of HIV-specific antibody responses in infants testing HIV-positive within 48 hours of birth and initiating early ART.

Secondary pathogenesis aims will test whether markers of neonatal immune quiescence are associated with the extent of seeding and rate of decline of the viral reservoir when ART is started at a young age and investigate whether markers in infant stool samples can be used as a non-invasive method of defining relevant immune and HIV-specific parameters associated with viral reservoir size.

The investigators hypothesize that developmental characteristics of newborn immunity may make this period the optimal time to begin ART and influence the seeding of the viral reservoir.

DETAILED DESCRIPTION:
Prevention of mother-to-child transmission (PMTCT) programs using antiretrovirals (ARVs) have had tremendous success in sub-Saharan Africa. However, HIV transmission continues to occur because (1) implementation of PMTCT is incomplete and (2) ARV interventions are not 100% effective in blocking infection. Thus the challenge of providing treatment to HIV-infected children is far from over. The capacity of early ART treatment to favorably influence the viral reservoir and potentially lead to post-treatment cessation viral control needs to be described in the population of infants, and to identify useful public health strategies.

ELIGIBILITY:
Inclusion Criteria:

* Point of care (POC) or laboratory-based test positive on a sample collected within 48 hours of birth.
* Mother willing and able to provide informed consent.

Exclusion Criteria:

* Expressed intention to leave the Johannesburg area permanently.
* Co-morbidities, birth defects or other conditions which in the opinion of the clinical team have a greater than 50% risk of mortality in the first days of life.
* Co-morbidities or conditions which in the opinion of the clinical team advise against initiation of ART within the first 48 hours of life.
* Active (uncontrolled) maternal psychiatric illness.

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Percent of patients with initial viral suppression | 24 weeks
  Suppression is defined as patients with plasma HIV RNA <50 copies/mL.

SECONDARY OUTCOMES:
Percent of patients maintaining viral suppression | Between 24 and104 weeks
  Suppression is defined as patients with plasma HIV RNA <50 copies/mL.
Prevalence of CD4 percentage greater than 30 | By 24 weeks and sustained through 104 weeks
  Patients that reached a normal CD4% level.
Prevalence of growth along curve within one standard deviation or upward trend | Up to 104 weeks
  By comparing viral growth curves.
Prevalence of detection of specific HIV antibody classes | 24 and 104 weeks
  HIV antibody detection
Size of the viral reservoir (copies/million cell) | Up to 104 weeks
  Quantification of viral reservoir

CONTACTS AND LOCATIONS:
Overall Officials: Louise Kuhn, PhD, Principal Investigator — Columbia University
Locations (1):
- Rahima Moosa Mother and Child Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Contact PI Non-identifying data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Based on availability of resources
Access Criteria: Scientific justification

REFERENCES:
- [Derived] Kuhn L, Paximadis M, Da Costa Dias B, Shen Y, Mncube S, Strehlau R, Shiau S, Patel F, Burke M, Technau KG, Sherman G, Loubser S, Abrams EJ, Tiemessen CT. Predictors of Cell-Associated Human Immunodeficiency Virus (HIV)-1 DNA Over 1 Year in Very Early Treated Infants. Clin Infect Dis. 2022 Mar 23;74(6):1047-1054. doi: 10.1093/cid/ciab586. PMID 34185838
- [Derived] Kuhn L, Strehlau R, Shiau S, Patel F, Shen Y, Technau KG, Burke M, Sherman G, Coovadia A, Aldrovandi GM, Hazra R, Tsai WY, Tiemessen CT, Abrams EJ; LEOPARD Study Team. Early antiretroviral treatment of infants to attain HIV remission. EClinicalMedicine. 2020 Jan 7;18:100241. doi: 10.1016/j.eclinm.2019.100241. eCollection 2020 Jan. PMID 31993578